CLINICAL TRIAL: NCT05083585
Title: A Randomized, Double-blind Phase 3 Study to Compare the Immunogenicity of Clinical Trial Material of an Ad26.RSV.preF-based Vaccine for Phase 3 With Clinical Trial Material Representative of Phase 2b in Adults Aged 60 to 75 Years
Brief Title: A Study Evaluating the Immunogenicity of Different Clinical Trial Materials of Ad26.RSV.preF- Based Vaccine in Adults Aged 60 - 75 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR109065; VAC18193RSV3004 (Other: Janssen Vaccines & Prevention B.V)
Record Dates: First submitted 2021-10-07; First posted 2021-10-19 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Virus Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Phase 3 Clinical Trial Material (CTM) (Experimental): Participants will receive a single intramuscular (IM) injection of adenovirus serotype 26 (Ad26). respiratory syncytial virus (RSV). prefusion conformation-stabilized F protein (preF)-based vaccine on Day 1, which is a Phase 3 CTM.
  Interventions: Biological: Ad26.RSV.preF-based vaccine
- Group 2: Phase 2b CTM (Experimental): Participants will receive a single IM injection of Ad26.RSV.preF-based vaccine on Day 1, which is a Phase 2b CTM.
  Interventions: Biological: Ad26.RSV.preF-based vaccine

INTERVENTIONS:
Biological: Ad26.RSV.preF-based vaccine — Ad26.RSV.preF-based vaccine will be administered as a single intramuscular injection.

SUMMARY:
The purpose of this study is to demonstrate non-inferiority in terms of humoral immune responses induced by vaccination with one dose of the Phase 3 clinical trial material (CTM) compared with one dose of the Phase 2b CTM.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to adhere to the prohibitions and restrictions specified in the protocol
* Before randomization, a participant must be postmenopausal (postmenopausal state is defined as no menses for 12 months without an alternative medical cause); and not intending to conceive by any methods
* In the investigator's clinical judgment, participant must be in stable health at the time of vaccination. Participants may have underlying illnesses such as hypertension, congestive heart failure, chronic obstructive pulmonary disease, type 2 diabetes, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms and signs are stable at the time of vaccination, and these conditions receive routine follow-up by the participant's healthcare provider. Participants will be included on the basis of medical history, and vital signs performed between informed consent form (ICF) signature and vaccination
* Must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study
* From the time of vaccination through 3 months after vaccination, agrees not to donate blood

Exclusion Criteria:

* Known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine)
* Abnormal function of the immune system resulting from clinical condition or medication
* History of acute polyneuropathy (example, Guillain-Barré syndrome) or chronic idiopathic demyelinating polyneuropathy
* History of thrombosis with thrombocytopenia syndrome (TTS) or heparin-induced thrombocytopenia and thrombosis (HITT)
* Has had major surgery (per the investigator's judgment) within 4 weeks before administration of the study vaccine or will not have recovered from surgery per the investigator's judgment at time of vaccination

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (9):
- United States (9):
  - Artemis Institute for Clinical Research, San Diego, California
  - Optimal Research, San Diego, California
  - Accel Research Sites, Lakeland, Florida
  - Optimal Research, Melbourne, Florida
  - Pharmax Research Clinic Inc, Miami, Florida
  - Research Institute of South Florida Inc, Miami, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridian Clinical Research, LLC, Cincinnati, Ohio
  - Tekton Research Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg: Participants received a single intramuscular (IM) injection of adenovirus serotype 26 pre-fusion conformation-stabilized F protein (Ad26.RSV.preF) 1.0*10^11 viral particles (vp) and respiratory syncytial virus prefusion F-protein (RSV preF) 150 micrograms (mcg) based vaccine mixture (Ad26/protein preF RSV) on Day 1, which was a representative of Phase 3 clinical trial material (CTM).
- Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg: Participants received a single IM injection of Ad26.RSV.preF 1.0*10^11 vp and RSV preF protein 150 mcg based vaccine mixture (Ad26/protein preF RSV) on Day 1, which was a representative of Phase 2b CTM.
Period: Overall Study
Arm/Group | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg
Started | 125 | 125
Vaccinated (Full Analysis Set [FAS]) | 123 | 125
Completed | 119 | 123
Not Completed | 6 | 2
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Randomized but not vaccinated | 2 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who received study vaccine, regardless of the occurrence of protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Total
Number analyzed (Participants) | 123 | 125 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (3.85) | 64.2 (4.34) | 64 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 63 | 128
  Male | 58 | 62 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 58 | 103
  Not Hispanic or Latino | 78 | 65 | 143
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 13 | 26
  White | 109 | 111 | 220
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 123 | 125 | 248

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Prefusion F-protein (preF) Antibodies as Assessed by Enzyme-linked Immunosorbent Assay (ELISA) 14 Days Post Vaccination
Description: GMTs of pre-F antibodies as assessed by ELISA at 14 days post administration of Ad26/protein preF RSV based vaccine were reported.
Time Frame: 14 days post vaccination on Day 1 (Day 15)
Population: The per-protocol immunogenicity (PPI) set included all randomized participants who received the study vaccine, and for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per liter (EU/L)
Arm/Group | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 114 | 120
ELISA units per liter (EU/L) | 5054 [4444 to 5748] | 4836 [4220 to 5543]

2. Secondary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) for 7 Days Post Vaccination
Description: Number of participants with solicited local AEs 7 days post vaccination on Day 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs were precisely defined events that participants were specifically asked about and which were noted by participants in the diary. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site).
Time Frame: Up to Day 7 post vaccination on Day 1 (up to Day 8)
Population: The full analysis set (FAS) included all participants who received study vaccination, regardless of the occurrence of protocol deviations. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 121 | 125
Participants | 84 | 74

3. Secondary Outcome: Number of Participants With Solicited Systemic AEs for 7 Days Post Vaccination
Description: Number of participants with solicited systemic AEs 7 days post vaccination on Day 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which were noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Up to Day 7 post vaccination on Day 1 (up to Day 8)
Population: The FAS included all participants who received study vaccination, regardless of the occurrence of protocol deviations. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 121 | 125
Participants | 76 | 77

4. Secondary Outcome: Number of Participants With Unsolicited AEs for 28 Days Post Vaccination
Description: Number of participants with unsolicited AEs 28 days post vaccination on Day 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant was not specifically questioned in the participant diary.
Time Frame: Up to Day 28 post vaccination on Day 1 (up to Day 29)
Population: The FAS included all participants who received study vaccination, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 123 | 125
Participants | 9 | 12

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) Until 6 Months Post Vaccination
Description: Number of participants with SAEs until 6 months post vaccination on Day 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: From Day 1 up to 6 months post vaccination on Day 1 (up to Day 183)
Population: The FAS included all participants who received study vaccination, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 123 | 125
Participants | 2 | 3

6. Secondary Outcome: Number of Participants With Adverse Event of Special Interests (AESIs) Until 6 Months Post Vaccination
Description: Number of participants with AESIs until 6 months post vaccination on Day 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Thrombosis with thrombocytopenia syndrome (TTS) was considered as an AESI.
Time Frame: From Day 1 up to 6 months post vaccination on Day 1 (up to Day 183)
Population: The FAS included all participants who received study vaccination, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 123 | 125
Participants | 0 | 0

7. Secondary Outcome: Respiratory Syncytial Virus (RSV) A2 Strain Neutralization Antibody Titers at 14 Days Post Vaccination
Description: RSV A2 strain neutralizing antibody titers of the vaccine-induced immune response was assessed through virus neutralization assay at 14 days post administration of Ad26/protein preF RSV based vaccine were expressed as 50 percent (%) inhibitory concentration (IC50) units.
Time Frame: 14 days post vaccination on Day 1 (Day 15)
Population: The PPI set included all randomized participants who received the study vaccine, and for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 114 | 120
Titers | 7710 [6623 to 8976] | 7256 [6231 to 8450]

ADVERSE EVENTS:
Time Frame: From Day 1 until 6 months post vaccination (up to Day 183)
Description: The full analysis set (FAS) included all participants who received study vaccine, regardless of the occurrence of protocol deviations.
Arm/Group | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg
All-Cause Mortality (participants affected / at risk) | 1/123 | 1/125
Serious Adverse Events (participants affected / at risk) | 2/123 | 3/125
Other Adverse Events (participants affected / at risk) | 3/123 | 2/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg (N=123) | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg (N=125)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Phase 3 CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg (N=123) | Group 2 (Phase 2b CTM): Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg (N=125)
Chills (General disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT05083585/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT05083585/SAP_001.pdf